CLINICAL TRIAL: NCT04035252
Title: Relation betwEen Abdominal Aorta and Carotid Artery Responses to SymPathetic stimulatiON uSing duplEx Ultrasound
Acronym: RESPONSE
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RESPONSE study
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Functional response; Abdominal aortic aneurysm; Carotid artery
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1. Young healthy group: Male or female between the age of 18 and 40 years old. No presence of systolic blood pressure >140 and/or diastolic blood pressure >90, cardiovascular history or antihypertensive medication
  Interventions: Diagnostic Test: Carotid artery reactivity test (CAR-test)
- 2. Patients with an AAA: Individuals (>60 years) with a small, stable, abdominal aortic aneurysm (i.e. AAA diameter of 30-50 mm)
  Interventions: Diagnostic Test: Carotid artery reactivity test (CAR-test)
- 3. Healthy older group: Healthy age- and sex- matched with group 2 with no presence of systolic blood pressure >140 and/or diastolic blood pressure >90, cardiovascular history or antihypertensive medication
  Interventions: Diagnostic Test: Carotid artery reactivity test (CAR-test)

INTERVENTIONS:
Diagnostic Test: Carotid artery reactivity test (CAR-test) — The CAR test will be applied to stimulate the sympathetic nervous system. This thermal stimulus is known to elevate blood pressure via sympathetic pathways, so it can be used to study the vascular response to sympathetic activation. The participant will submerge their left hand in a bucket of ice water (approximately 4 degrees celcius) for 3 minutes, which is reported to be sufficient to induce a maximal dilation in the common carotid artery. At baseline and every minute after the hand is submerged in ice water, the blood pressure will be measured to check whether a sympathetic stimulation is achieved. During this test as well the carotid artery as the abdominal aorta will be visualized using ultrasound.

SUMMARY:
Abdominal aortic aneurysm (AAA) is a common vascular disease and associated with risk of rupture, but also with a high cardiovascular (CV) event rate. A key difficulty in AAA is predicting these life-threatening complications. Recent studies suggest that the endothelial function of the abdominal aorta might have a correlation with the disease development. A novel, easy to perform, non-invasive test can assess central artery endothelial function (i.e. the carotid artery reactivity (CAR)). The CAR test is based on the cold pressure test (CPT), which induces sympathetic stimulation by placing one hand in cold water. Using duplex ultrasound, central artery blood flow and diameter responses can be examined.

Previous work has demonstrated that the CPT is associated with an increase in abdominal aortic diameter, whilst others found that the carotid and coronary artery diameter also shows dilation. Interestingly, a previous study found a strong correlation between carotid and coronary artery diameter responses to the CPT, whilst these artery responses show independent prognostic value for future cardiovascular events in patients with peripheral arterial disease. Possibly, similarity may be present in central artery reactivity to the CPT. To date, no study examined whether carotid and aorta responses are in agreement during the CPT. Given the potential importance of central artery vasoreactivity for AAA, the CAR-test may have potential in this group, especially given the relative simplicity of measuring the carotid artery.

The aim of this explorative study is to investigate the correlation between the magnitude of the abdominal aorta and the carotid artery diameter and blood flow responses during the sympathetic stimulation (using the cold pressor test) between healthy young, healthy older and individuals with AAA.

DETAILED DESCRIPTION:
The present study is an explorative, observational study, which will include in total 60 participants divided over 3 groups; healthy young adults, healthy older adults and patients with a stable abdominal aortic aneurysm (i.e. 30-50 mm), who are currently under threshold for repair. When participants meet the criteria, they will be informed about the study and they will be asked for their written informed consent, when they are willing to participate. Every participant only need to visit one time, which takes approximately 30 minutes. Participant characteristics will be registered, including traditional risk factors and CV history. Subsequently, the investigators will perform the CAR-test, which takes approximately 15 minutes. Prior to the CAR-test, participants should follow some instructions with regard to food and fluid intake according to a physiological guideline, which can influence this test.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy group: Male or female between the age of 18 and 40 years old;
* Older healthy group: Male or female, which are age-/sex-matched with the AAA patients group;
* AAA patients group: Male or female with an abdominal aortic aneurysm who is still under surveillance, with a diameter between 3.0 and 5.0 cm and at least 18 years old. These patients may participate in the 1-2-3 Trial, which is a similar approved investigation by CMO region Arnhem-Nijmegen with registration number 2019-5216.
* Informed consent form understood and signed;

Exclusion Criteria:

* Psychiatric or other conditions that may interfere with the study;
* Participating in another clinical study, interfering on outcomes;
* With regard to the necessary quality of the ultrasound images, BMI ≥ 30 kg/m2;
* Increased risk for coronary spasms (score Rose-questionnaire ≥2; this questionnaire can be found in the Appendix);
* Known carotid artery disease
* Presence of Raynaud's phenomenon, Marfan syndrome, chronic pain syndrome at upper extremity(s), presence of an AV fistula or shunt, open wounds to the upper extremity(s), and/or scleroderma associated with placing the hand in ice water;
* Recent (<3 months) presence of angina pectoris, myocardial infarction, cerebral infarction, and/or heart failure, or PAD treatment.
* Healthy groups:

  * Systolic blood pressure >140 and/or diastolic blood pressure >90
  * Cardiovascular history
  * Antihypertensive medication

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. twenty healthy, young (18-40 years) subjects,
  2. twenty older subjects (>60 years) with a small, stable abdominal aortic aneurysm (i.e. AAA diameter of 30-50 mm), and
  3. twenty healthy, age-/sex matched with group 2. We aim to include an equal number of male and females in both groups.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
CAR-test | Baseline
  Percentage of vasodilation/vasoconstriction to the CAR test at the common carotid artery
CAR-test | Baseline
  Percentage of vasodilation/vasoconstriction to the CAR test at the abdominal aorta

SECONDARY OUTCOMES:
CAR-test | Baseline
  Magnitude of the blood flow and perfusion response of the carotid artery
CAR-test | Baseline
  Timing of the blood flow and perfusion response of the carotid artery
CAR-test | Baseline
  Magnitude of the blood flow and perfusion response of the abdominal aorta
CAR-test | Baseline
  Timing of the blood flow and perfusion response of the abdominal aorta
CAR-test | Baseline
  Blood pressure response
CAR-test | Baseline
  Heart rate response
Age | Baseline
  Age

OTHER OUTCOMES:
Demographic characteristics | Baseline
  Gender
Demographic characteristics | Baseline
  If current smoker
Demographic characteristics | Baseline
  Height
Demographic characteristics | Baseline
  Weight
Demographic characteristics | Baseline
  Medical history
Demographic characteristics | Baseline
  Blood pressure
Demographic characteristics | Baseline
  Heart rate
Medication use | Baseline
  Ask about: Statins
Medication use | Baseline
  Ask about: Beta-blockers
Medication use | Baseline
  Ask about: Sympathicomimetica
Medication use | Baseline
  Ask about: Anti-platelets
Medication use | Baseline
  Ask about: Anti-coagulants
Medication use | Baseline
  Ask about: Anti-hypertensives (questioned)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, MD, Prof, Principal Investigator — Rijnstate Hospital
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Radboudumc, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: Undecided